CLINICAL TRIAL: NCT03563976
Title: Multi Parametric Image Analysis and Correlation With Outcomes in Lung Cancer Screening and Early Stage Lung Cancer
Brief Title: Multiparametric Image Analysis and Correlation With Outcomes in Lung Cancer Screening and Early Stage Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Jing Wang, Associate Professor of Medicine, University of Texas Southwestern Medical Center
Other Study IDs: STU 122014-052
Record Dates: First submitted 2018-05-18; First posted 2018-06-20 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Lung Cancer
Keywords: Early Stage Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Retrospective Studies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Retrospective Study — The medical charts are the subjects. The institutional charts will be identified by the use of definitive radiation therapy correlating with an early stage lung cancer diagnosis during the above time frame. The data from these charts will be entered into a password protected excel spreadsheet. The charts will be identified by name, medical record number, date of birth, and social security number. These are all patients treated by all hospitals and clinics affiliated with UTSW and Parkland. At the time of study, some of the patients will have expired but some will be alive and in the regional North Texas area. Thus, given the minimal risk nature of this retrospective chart review, we could not reasonably conduct this research with a full waiver of consent. The NLST external dataset is proved by the NCI, with no identifying characteristics.

SUMMARY:
Determine whether CT-based multiparametric analytical models may improve prediction of biopsy and treatment outcome in patients undergoing screening CT scan and/or treatment for early stage lung cancer

DETAILED DESCRIPTION:
The hypothesis is that multiparametric models that incorporate complex image information from screening CT scans will improve prediction of the outcome of subsequent lung biopsy, an invasive diagnostic procedure. In this project, we will construct an image feature-based multiparametric prognostic model for biopsy outcome from screening lung CT scans performed at our institution, and then validate it using theNLST imaging and clinical outcomes dataset.

This study involves no treatment or invasive procedures. Investigator will review all charts of patients who were treated for early stage lung cancer with definitive radiation therapy at UTSW or Parkland Memorial hospital, diagnosed with a malignancy from January 1, 2004 to October 31, 2014, to compile demographic, diagnostic, therapeutic, outcome, and toxicity data. Investigator expect that this will include approximately 200 patient charts. This data will be analyzed statistically and used for future directed research. Investigator will also analyze an anonymized dataset of patients from the National Lung Cancer Screening Trial (NLST) provided by the National Cancer Institute (NCI)

ELIGIBILITY:
Inclusion Criteria:

Patients that have been diagnosed with lung cancer, and are treated at Department of Radiation Oncology, UTSW or Parkland Memorial Hospital.

Exclusion Criteria:

There will be no absolute exclusion criteria as long as the inclusion criteria have been met.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The medical charts are the subjects. Risk will be minimized by protecting patient data through the use of de-identification of patient identifiers and password protected data collection. The information will be given only to faculty members and statisticians involved in the research project. The data will be disclosed only for analytical purposes.
  Confidentiality will be maintained by adhering to HIPAA guidelines. The location of the data will be maintained at the worksite of the PI and the research coordinator in the Moncrief Radiation Oncology Department on the North Campus at UTSW. Risks will be minimized by protecting patient data and using it only for research purposes for retrospective analysis.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2015-02-18 (Actual); Primary Completion 2026-03-20 (Estimated); Study Completion 2028-03-15 (Estimated)

PRIMARY OUTCOMES:
Determine whether CT-based multiparametric analytical models may improve prediction of biopsy and treatment outcome in patients undergoing screening CT scan and/or treatment for early stage lung cancer | 10 years
  We will review all charts of patients who were treated for early stage lung cancer with definitive radiation therapy at UTSW or Parkland Memorial hospital, diagnosed with a malignancy from January 1, 2004 to October 31, 2014, to compile demographic, diagnostic, therapeutic, outcome, and toxicity data. The data will be subject to standard descriptive, parametric, and nonparametric hypothesis testing with biostatistical analyses. We will also analyze an anonymized dataset of patients from the National Lung Cancer Screening Trial (NLST) provided by the National Cancer Institute (NCI) including screening images and diagnostic outcomes to validate models generated using institutional data.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Wang, MD, Principal Investigator — UTSW Radiation Oncology
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided